CLINICAL TRIAL: NCT02370602
Title: An Open-Label [^11C]T-773 Positron Emission Tomography Study to Determine Phosphodiesterase10A Occupancy by TAK-063 After a Single Oral Dose in Human Volunteers
Brief Title: An [^11C]T-773 Positron Emission Tomography (PET) Study to Determine Phosphodiesterase10A Occupancy by TAK-063
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAK-063_103; U1111-1165-3362 (Registry Identifier: WHO); 2012-004576-18 (EudraCT Number)
Record Dates: First submitted 2015-02-18; First posted 2015-02-25 (Estimated); Results first posted 2015-03-20 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy
MeSH Terms: interventions — 1-(2-fluoro-4-(1H-pyrazol-1-yl)phenyl)-5-methoxy-3-(1-phenyl-1H-pyrazol-5-yl)pyridazin-4(1H)-one; T-773 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pilot Cohort: [^11C]T-773 + TAK-063 (Experimental): [^11C]T-773 <8 μg; 400MBq ± 10%, intravenous (IV), once on Days 1 and 2 prior to PET scans and TAK-063 30 mg or 1000 mg, tablets, orally, once on Day 2 and after PET scan #2 and prior to PET scan #3 and [^11C]T-773 IV after TAK-063 and prior to PET scan #3 on Day 2.
  Interventions: Drug: TAK-063; Drug: [^11C]T-773
- Main Cohort: TAK-063 + [^11C]T-773 (Experimental): TAK-063 3 to 100 mg, tablets, orally, once, on Day 1, and [^11C]T-773 <8 μg; 400MBq ± 10%, intravenously (IV), prior to PET scans, twice on Day 1 (before and after administration of TAK-063) and once on Day 2 .
  Interventions: Drug: TAK-063; Drug: [^11C]T-773

INTERVENTIONS:
Drug: TAK-063 — TAK-063 tablets
Drug: [^11C]T-773 — [^11C]T-773 IV solution

SUMMARY:
The purpose of this study is to estimate phosphodiesterase 10A (PDE10A) occupancy in brain following a single dose of TAK-063.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-063. TAK-063 is was tested to estimate phosphodiesterase10A (PDE10A) occupancy in the brain following a single dose of TAK-063. This study used positron emission tomography (PET) scans to look at changes in the volume of tissue distribution before and after TAK-063 administration to calculate PDE10A occupancy in the brain.

The study enrolled 13 participants. Participants were assigned to a treatment group based on an enrollment schedule. The first 4 participants were assigned to the Pilot Cohort and received one dose of TAK-063 30 mg or 1000 mg tablets. The remaining participants were enrolled into the Main Cohort and received one dose of TAK-063 at 3, 10, 30 or 100 mg. Participants in both cohorts also received 3 separate intravenous infusions of [^11C]T-773 <8 μg; 400MBq ± 10% followed by a PET scan.

This single-centre trial was conducted in Sweden. The overall time to participate in this study was 46 days. Participants made 3 visits to the clinic, including one 3-day period of confinement to the clinic. Participants were contacted by phone on Day 16 for follow-up safety assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Has never previously participated in a positron emission tomography (PET) study (lifetime).
2. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
3. The participant, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
4. Is a healthy adult male, as determined by a physician based upon medical history and physical examination findings at Screening.
5. Is aged 20 to 45 years, inclusive, at the time of informed consent.
6. Weighs at least 50 kg and less than 100 kg and has a body mass index (BMI) between 18 and 32 kg/m^2 inclusive at Screening.
7. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after last dose.
8. Has clinical laboratory evaluations (including clinical chemistry, hematology and complete urinalysis) within the reference range for the testing laboratory, unless the results are deemed not to be clinically significant (CS) by the investigator or sponsor at screening. Participants must have normal hemoglobin levels.
9. Has a normal magnetic resonance imaging (MRI) scan or findings that are deemed not clinically significant at screening (the MRI scan may be performed on a day after other screening activities have been performed but before dosing).

Exclusion Criteria:

1. Has received any investigational compound within 90 days prior to Screening.
2. Has received TAK-063 in a previous clinical study or as a therapeutic agent.
3. Is an immediate family member, study site employee, or in a dependant relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
4. Has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, endocrine disease, or psychiatric disorder, or other abnormality, which may impact the ability of the participant to participate or potentially confound the study results.
5. Has a known hypersensitivity to any component of the formulation of TAK-063 or [^11C]T-773.
6. Has a positive urine drug result for drugs of abuse or a positive breathalyzer test for alcohol at Screening or Day -1.
7. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the screening visit or is unwilling to agree to abstain from alcohol until discharge from the Phase 1 unit and drugs throughout the study.
8. Has taken any excluded medication, supplements, or food products listed in the Excluded Medications and Dietary Products table.
9. Intends to donate sperm during the course of the study or within 12 weeks after last dose.
10. Has evidence of current cardiovascular, central nervous system, hepatic, hematopoietic disease, renal dysfunction, metabolic or endocrine dysfunction, serious allergy, asthma hypoxemia, hypertension, seizures, or allergic skin rash. There is any finding in the participant's medical history, physical examination, or safety laboratory tests giving reasonable suspicion of a disease that would contraindicate taking TAK-063 or a similar drug in the same class, or that might interfere with the conduct of the study. This includes, but is not limited to, peptic ulcer disease, seizure disorders, and cardiac arrhythmias.
11. The participant, in the opinion of the investigator, has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (ie, a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis frequent [more than once per week] occurrence of heartburn, or any surgical intervention [eg, cholecystectomy]).
12. Has a history of cancer, except basal cell carcinoma which has been in remission for at least 5 years prior to Day 1.
13. Has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV), human immunodeficiency virus (HIV) antibody/antigen, at Screening.
14. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 28 days prior to Check-In Day -1.
15. Has poor peripheral arterial/venous access or recent arm or wrist trauma.
16. Has donated or lost 450 mL or more of his blood volume (including plasmapheresis), or had a transfusion of any blood product within 3 months prior to Day 1.
17. Has a Screening or Check-in (Day -1) abnormal (clinically significant) electrocardiogram (ECG).
18. Has a supine blood pressure outside the ranges of 90 to 140 mm Hg for systolic and 50 to 90 mm Hg for diastolic, if out of range may be repeated once for eligibility determination within a maximum of 5 minutes, at the Screening Visit or Check-in (Day -1).
19. Has a resting heart rate outside the range 45 to 90 beats per minute (bpm), if out of range may be repeated once for eligibility determination within a maximum of 5 minutes, at the Screening Visit or Check-in (Day -1).
20. Has an increase in pulse of ≥30 beats per minute or an increase in pulse ≥120 beats per minute within 3 minutes of standing at Screening.
21. Has a decrease of ≥20 mm Hg in systolic blood pressure or a decrease of ≥10 mm Hg in diastolic blood pressure within 3 minutes of standing at Screening.
22. Has a QT interval with Fridericia correction method (QTcF) >430 ms or PQ interval outside the range 120 to 220 ms, if out of range may be repeated once for eligibility determination within a maximum of 5 minutes, at the Screening Visit or Check-in (Day -1) Visit.
23. Has abnormal Screening laboratory values that suggest a clinically significant underlying disease or participant with the following lab abnormalities: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >1.5 the upper limits of normal.
24. Has had administration of radioactive substances or exposure to significant radiation (eg, serial x-ray or computed tomography [CT] scans, barium meal) within the past 12 months prior to Day 1 predose.
25. Has any condition that would prevent an MRI from accurately or safely being performed (eg, claustrophobia, cardiac pacemaker, metallic implants or clips)
26. Has any condition that would prevent the performance of a safe or accurate PET scan.
27. Has any clinically significant MRI finding that in the opinion of the investigator would exclude the participant.
28. Is unwilling to refrain from strenuous exercise from 120 hours before Check-in (Day -1) until discharge from the Phase 1 unit.
29. Has a risk of suicide according to the Investigator's clinical judgment (eg, per Columbia-Suicide Severity Rating Scale (C-SSRS) or has made a suicide attempt in the previous 6 months.
30. Has abnormal international normalized ratio (INR) or activated prothrombin time (aPTT) or other risk of bleeding disorder.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Sweden from 13 August 2013 to 12 March 2014.
Pre-assignment Details: Healthy Volunteers received 1 of 5 treatments: 11C T-773,Tak-063 3 mg, Tak-063 10 mg, Tak-063 30 mg, Tak-063 100 mg or Tak-063 1000 mg.
Groups:
- [^11C]T-773 Only: [^11C]T-773 <8 μg; 400MBq ± 10%, intravenous (IV), once on Days 1 and 2 only.
- TAK-063 3 mg + [^11C]T-773: TAK-063 3 mg, tablets, orally, once, on Day 1, and [^11C]T-773 <8 μg; 400MBq ± 10%, intravenously (IV), prior to PET scans, twice on Day 1 (before and after administration of TAK-063) and once on Day 2.
- TAK-063 10 mg + [^11C]T-773: TAK-063 10 mg, tablets, orally, once, on Day 1, and [^11C]T-773 <8 μg; 400MBq ± 10%, intravenously (IV), prior to PET scans, twice on Day 1 (before and after administration of TAK-063) and once on Day 2.
- TAK-063 30 mg + [^11C]T-773: For main cohort, TAK-063 30 mg, tablets, orally, once, on Day 1, and [^11C]T-773 <8 μg; 400MBq ± 10%, intravenously (IV), prior to PET scans, twice on Day 1 (before and after administration of TAK-063) and once on Day 2. For pilot cohort, TAK-063 30 mg, tablets, orally, once on Day 2, and [^11C]T-773 <8 μg; 400MBq ± 10%, intravenously (IV), prior to PET scans, once on Day 1 (before and after administration of TAK-063) and twice on Day 2.
- TAK-063 100 mg + [^11C]T-773: TAK-063 100 mg, tablets, orally, once, on Day 1, and [^11C]T-773 <8 μg; 400MBq ± 10%, intravenously (IV), prior to PET scans, twice on Day 1 (before and after administration of TAK-063) and once on Day 2.
- TAK-063 1000 mg + [^11C]T-773: TAK-063 1000 mg, tablets, orally, once, on Day 2, and [^11C]T-773 <8 μg; 400MBq ± 10%, intravenously (IV), prior to PET scans, once on Day 1 and twice on Day 2 (before and after administration of TAK-063).
Period: Overall Study
Arm/Group | [^11C]T-773 Only | TAK-063 3 mg + [^11C]T-773 | TAK-063 10 mg + [^11C]T-773 | TAK-063 30 mg + [^11C]T-773 | TAK-063 100 mg + [^11C]T-773 | TAK-063 1000 mg + [^11C]T-773
Started | 1 | 2 | 2 | 3 | 3 | 2
Completed | 0 | 2 | 2 | 3 | 3 | 2
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Pretreatment Event/Adverse Event | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- [^11C]T-773: [^11C]T-773 <8 μg; 400MBq ± 10%, intravenous (IV), once on Days 1 and 2 only.
- Total: Total of all reporting groups
Arm/Group | [^11C]T-773 | TAK-063 3 mg + [^11C]T-773 | TAK-063 10 mg + [^11C]T-773 | TAK-063 30 mg + [^11C]T-773 | TAK-063 100 mg + [^11C]T-773 | TAK-063 1000 mg + [^11C]T-773 | Total
Number analyzed (Participants) | 1 | 2 | 2 | 3 | 3 | 2 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.0 (NA) — Standard deviation can not be calculated for 1 participant. | 27.5 (4.95) | 26.5 (0.71) | 37.7 (7.09) | 26.7 (3.51) | 27.0 (1.41) | 29.2 (6.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 1 | 2 | 2 | 3 | 3 | 2 | 13
Race/Ethnicity, Customized [Number; unit: participants]
  White | 1 | 2 | 2 | 3 | 3 | 2 | 13
Region of Enrollment [Number; unit: participants]
  Sweden | 1 | 2 | 2 | 3 | 3 | 2 | 13
Height [Mean (Standard Deviation); unit: cm] | 183.0 (NA) — Standard deviation can not be calculated for 1 participant. | 180.5 (4.95) | 180.0 (1.41) | 178.0 (8.19) | 179.3 (7.51) | 177.0 (4.24) | 179.2 (5.20)
Weight [Mean (Standard Deviation); unit: kg] | 83.00 (NA) — Standard deviation can not be calculated for 1 participant. | 76.40 (0.566) | 90.50 (4.950) | 85.90 (3.651) | 83.27 (15.938) | 80.65 (4.596) | 83.51 (8.233)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.78 (NA) — Standard deviation can not be calculated for 1 participant. | 23.47 (1.117) | 27.92 (1.089) | 27.27 (3.267) | 25.86 (4.584) | 25.80 (2.701) | 26.04 (2.883)
Smoking Classification [Number; unit: participants]
  Never smoked | 1 | 2 | 2 | 1 | 3 | 2 | 11
  Current smoker | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ex-smoker | 0 | 0 | 0 | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Phosphodiesterase 10A (PDE10A) Occupancy of Brain Regions With [^11C]T-773 at 3 Hours Following a Single Dose of TAK-063
Description: Volume of tissue distribution (Vt) values will be estimated by several quantitative methods for each positron emission tomography (PET) scan. Based on the change in Vt before and after TAK-063 administration, PDE10A occupancy will be calculated. PET scan #2 in the Pilot Cohort and PET scan #1 in the Main Cohort will be used as a baseline for the occupancy calculation. Occupancy is reported for putamen only.
Time Frame: 3 hours post-dose
Population: Pharmacodynamic Analysis Set includes all participants with data available for pharmacodynamic analysis..
Measure: Mean (Standard Deviation); unit: Percent
Groups:
- TAK-063 10 mg: TAK-063 10 mg, tablets, orally, once, on Day 1, and [^11C]T-773 <8 μg; 400MBq ± 10%, intravenously (IV), prior to PET scans, twice on Day 1 (before and after administration of TAK-063) and once on Day 2.
Arm/Group | TAK-063 3 mg + [^11C]T-773 | TAK-063 10 mg | TAK-063 30 mg + [^11C]T-773 | TAK-063 100 mg + [^11C]T-773 | TAK-063 1000 mg + [^11C]T-773
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 2
Percent | 14.400 (16.4049) | 26.650 (2.4749) | 39.333 (11.1096) | 53.633 (0.9074) | 69.350 (3.8891)

2. Secondary Outcome: Phosphodiesterase 10A (PDE10A) Occupancy of Brain Regions With [^11C]T-773 at 23 Hours Following a Single Dose of TAK-063
Description: Volume of tissue distribution (Vt) values will be estimated by several quantitative methods for each positron emission tomography (PET) scan. Based on the change in Vt before and after TAK-063 administration, PDE10A occupancy will be calculated. PET scan #2 in the Pilot Cohort and PET scan #1 in the Main Cohort will be used as a baseline for the occupancy calculation. Data was not available for participants in the pilot cohort. Occupancy is reported for putamen only.
Time Frame: 23 hours post-dose
Population: Pharmacodynamic Analysis Set includes all participants with data available for pharmacodynamic analysis.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | TAK-063 3 mg + [^11C]T-773 | TAK-063 10 mg + [^11C]T-773 | TAK-063 30 mg + [^11C]T-773 | TAK-063 100 mg + [^11C]T-773
Number analyzed (Participants) | 2 | 2 | 1 | 3
Percent | -2.250 (0.7778) | 14.750 (1.7678) | 18.800 (NA) — Standard deviation can not be calculated for 1 participant. | 24.167 (18.6001)

3. Secondary Outcome: Percentage of Participants Who Experienced at Least 1 Treatment-Emergent Adverse Event
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: First dose of study drug to 30 days after last dose of study drug (up to 46 days)
Population: Safety analysis set included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- TAK-063: TAK-063 3 to 1000 mg, tablets, orally, once, on Day 1.
Arm/Group | [^11C]T-773 | TAK-063
Number analyzed (Participants) | 13 | 12
percentage of participants | 38.5 | 75.0

4. Secondary Outcome: Percentage of Participants With Markedly Abnormal Safety Laboratory Findings
Description: The percentage of participants with any markedly abnormal standard safety laboratory values was collected throughout study.
Time Frame: From Day 1 to Day 16
Population: Safety analysis set included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | [^11C]T-773 | TAK-063 3 mg + [^11C]T-773 | TAK-063 10 mg + [^11C]T-773 | TAK-063 30 mg + [^11C]T-773 | TAK-063 100 mg + [^11C]T-773 | TAK-063 1000 mg + [^11C]T-773
Number analyzed (Participants) | 13 | 2 | 2 | 3 | 3 | 2
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants With Markedly Abnormal Vital Sign Measurements
Description: The percentage of participants with any markedly abnormal standard vital sign measurements was collected throughout study. BL=baseline. bpm=beats per minute.
Time Frame: From Day 1 to Day 16
Population: Safety analysis set included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | [^11C]T-773 | TAK-063 3 mg + [^11C]T-773 | TAK-063 10 mg + [^11C]T-773 | TAK-063 30 mg + [^11C]T-773 | TAK-063 100 mg + [^11C]T-773 | TAK-063 1000 mg + [^11C]T-773
Number analyzed (Participants) | 13 | 2 | 2 | 3 | 3 | 2
percentage of participants
  During Treatment (tx) - >Upper Cut-off | 0 | 0 | 0 | 0 | 0 | 0
  During tx - <Lower Cut-off | 38.5 | 50.0 | 50.0 | 33.3 | 66.7 | 0
  During tx - Change Relative to BL Upper Criteria | 7.7 | 0 | 0 | 0 | 0 | 50.0
  During tx - Change Relative to BL Lower Criteria | 0 | 0 | 50.0 | 0 | 0 | 0
  During tx - Overall | 46.2 | 50.0 | 100.0 | 33.3 | 66.7 | 50.0
  Pulse (bpm) - >120 bpm | 0 | 0 | 0 | 0 | 0 | 0
  Pulse (bpm) - <50 bpm | 30.8 | 50.0 | 50.0 | 33.3 | 66.7 | 0
  Pulse (bpm) - Increase of >30 bpm | 0 | 0 | 0 | 0 | 0 | 0
  Pulse (bpm) - Decrease of >30 bpm | 0 | 0 | 0 | 0 | 0 | 0
  Pulse (bpm) - Overall | 30.8 | 50.0 | 50.0 | 33.3 | 66.7 | 0
  Systolic Blood Pressure (mmHg) - >180 mmHg | 0 | 0 | 0 | 0 | 0 | 0
  Systolic Blood Pressure (mmHg) - <85 mmHg | 0 | 0 | 0 | 0 | 0 | 0
  Systolic Blood Pressure - Increase of >40 mmHg | 0 | 0 | 0 | 0 | 0 | 0
  Systolic Blood Pressure - Decrease of >40 mmHg | 0 | 0 | 0 | 0 | 0 | 0
  Systolic Blood Pressure (mmHg) - Overall | 0 | 0 | 0 | 0 | 0 | 0
  Diastolic Blood Pressure (mmHg) - >110 mmHg | 0 | 0 | 0 | 0 | 0 | 0
  Diastolic Blood Pressure (mmHg) - <50 mmHg | 0 | 0 | 0 | 0 | 0 | 0
  Diastolic BP (mmHg) - Increase of >20 mmHg | 7.7 | 0 | 0 | 0 | 0 | 50.0
  Diastolic BP (mmHg) - Decrease of >20 mmHg | 0 | 0 | 50.0 | 0 | 0 | 0
  Diastolic Blood Pressure (mmHg) - Overall | 7.7 | 0 | 50.0 | 0 | 0 | 50.0
  Temperature (Degree C) - >37.7 C | 0 | 0 | 0 | 0 | 0 | 0
  Temperature (Degree C) - <35.6 C | 7.7 | 50.0 | 0 | 0 | 0 | 0
  Temperature (Degree C) - Overall | 7.7 | 50.0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants With Markedly Abnormal Criteria for Safety Electrocardiogram (ECG) Parameters
Description: The percentage of participants with any markedly abnormal standard 12-lead ECG measurements.
  QTc - Bazett's Interval (msec) is ≥500 msec OR ≥30 msec change from Baseline and ≥450 msec
Time Frame: From Day 1 to Day 16
Population: Safety analysis set included all participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | [^11C]T-773 | TAK-063 3 mg + [^11C]T-773 | TAK-063 10 mg + [^11C]T-773 | TAK-063 30 mg + [^11C]T-773 | TAK-063 100 mg + [^11C]T-773 | TAK-063 1000 mg + [^11C]T-773
Number analyzed (Participants) | 13 | 2 | 2 | 3 | 3 | 2
percentage of participants
  Heart Rate (bpm) - <50 bpm | 7.7 | 50.0 | 50.0 | 33.3 | 66.7 | 0
  Heart Rate (bpm) - Overall | 7.7 | 50.0 | 50.0 | 33.3 | 66.7 | 0
  RR Interval (msec) - ≥1440 msec | 0 | 0 | 0 | 33.3 | 0 | 0
  RR Interval (msec) - ≤600 msec | 0 | 0 | 0 | 0 | 0 | 0
  RR Interval (msec) - Overall | 0 | 0 | 0 | 33.3 | 0 | 0
  PR Interval (msec) - ≥200 msec | 0 | 0 | 0 | 33.3 | 0 | 0
  PR Interval (msec) - ≤80 msec | 0 | 0 | 0 | 0 | 0 | 0
  PR Interval (msec) - Overall | 0 | 0 | 0 | 33.3 | 0 | 0
  QRS Interval (msec) - ≥180 msec | 0 | 0 | 0 | 0 | 0 | 0
  QRS Interval (msec) - ≤80 msec | 0 | 0 | 0 | 0 | 0 | 0
  QRS Interval (msec) - Overall | 0 | 0 | 0 | 0 | 0 | 0
  QT Interval (msec) - ≥460 msec | 0 | 0 | 0 | 33.3 | 0 | 0
  QT Interval (msec) - <280 msec | 0 | 0 | 0 | 0 | 0 | 0
  QT Interval (msec) - Overall | 0 | 0 | 0 | 33.3 | 0 | 0
  QTc - Bazett's Interval (msec) - Overall | 0 | 0 | 0 | 0 | 0 | 0
  QTc - Fredericia's Interval (msec) - Overall | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-063 and TAK-063 Metabolite M-I
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: Pilot Cohort: Day 2 predose and at multiple time points (up to 24 hours) post-dose. Main Cohort: Day 1 predose and at multiple time points (up to 24 hours) post-dose.
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TAK-063 3 mg + [^11C]T-773 | TAK-063 10 mg + [^11C]T-773 | TAK-063 30 mg + [^11C]T-773 | TAK-063 100 mg + [^11C]T-773 | TAK-063 1000 mg + [^11C]T-773
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 2
ng/mL
  TAK-063 | 11.25 (3.323) | 22.78 (0.035) | 80.67 (35.147) | 77.05 (16.898) | 258.75 (18.031)
  TAK-063 Metabolite M-I | 15.60 (7.637) | 19.65 (0.283) | 49.63 (18.393) | 80.43 (26.831) | 146.50 (10.607)

8. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-063 and TAK-063 Metabolite M-I
Description: Time to reach the maximum plasma concentration (Cmax), equal to time (hours) to Cmax.
Time Frame: as for outcome 7
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | TAK-063 3 mg + [^11C]T-773 | TAK-063 10 mg + [^11C]T-773 | TAK-063 30 mg + [^11C]T-773 | TAK-063 100 mg + [^11C]T-773 | TAK-063 1000 mg + [^11C]T-773
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 2
hour
  TAK-063 | 1.25 (0.354) | 2.99 (0.018) | 1.33 (0.289) | 2.33 (0.563) | 2.25 (1.137)
  TAK-063 Metabolite M-I | 1.50 (0.000) | 2.99 (0.018) | 1.64 (1.116) | 2.00 (0.000) | 2.79 (1.120)

9. Secondary Outcome: AUC(0-tlqc): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-063 and TAK-063 Metabolite M-I
Description: (AUC(0-tlqc) is a measure of total plasma exposure to the drug from Time 0 to Time of the Last Quantifiable Concentration (AUC[0-tlqc]).
Time Frame: as for outcome 7
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | TAK-063 3 mg + [^11C]T-773 | TAK-063 10 mg + [^11C]T-773 | TAK-063 30 mg + [^11C]T-773 | TAK-063 100 mg + [^11C]T-773 | TAK-063 1000 mg + [^11C]T-773
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 2
ng*hr/mL
  TAK-063 | 91.42 (5.795) | 318.56 (66.183) | 774.76 (127.644) | 897.17 (181.699) | 3288.62 (109.282)
  TAK-063 Metabolite M-I | 88.74 (23.833) | 245.24 (30.128) | 519.92 (233.914) | 850.26 (325.161) | 1859.28 (308.436)

10. Secondary Outcome: AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours Postdose for TAK-063 and TAK-063 Metabolite M-I
Description: AUC(0-24) is a measure of total plasma exposure to the drug from Time 0 to 24 hours post-dose.
Time Frame: as for outcome 7
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | TAK-063 3 mg + [^11C]T-773 | TAK-063 10 mg + [^11C]T-773 | TAK-063 30 mg + [^11C]T-773 | TAK-063 100 mg + [^11C]T-773 | TAK-063 1000 mg + [^11C]T-773
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 2
ng*hr/mL
  TAK-063 | 92.55 (5.348) | 324.98 (68.303) | 774.44 (129.997) | 910.12 (184.418) | 3289.62 (110.695)
  TAK-063 Metabolite M-I | 89.64 (23.672) | 249.82 (31.357) | 519.82 (233.869) | 864.14 (332.414) | 1859.97 (309.411)

11. Secondary Outcome: Average Plasma Concentration on Day 1 (Cavg) for TAK-063 and TAK-063 Metabolite M-I
Description: Cavg is the average plasma concentration on Day 1, calculated as AUC(0-24)/24.
Time Frame: as for outcome 7
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TAK-063 3 mg + [^11C]T-773 | TAK-063 10 mg + [^11C]T-773 | TAK-063 30 mg + [^11C]T-773 | TAK-063 100 mg + [^11C]T-773 | TAK-063 1000 mg + [^11C]T-773
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 2
ng/mL
  TAK-063 | 3.86 (0.223) | 13.54 (2.846) | 32.27 (5.417) | 37.92 (7.684) | 137.07 (4.612)
  TAK-063 Metabolite M-I | 3.74 (0.986) | 10.41 (1.307) | 21.66 (9.745) | 36.01 (13.851) | 77.50 (12.892)

12. Secondary Outcome: CL/F: Oral Clearance of TAK-063
Description: CL/F is apparent clearance of the drug from the plasma, calculated as the drug dose divided by area under the curve from time 0 to 24 hours post-dose, after multiple dosing (at steady state).
Time Frame: as for outcome 7
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: liter/hour
Arm/Group | TAK-063 3 mg + [^11C]T-773 | TAK-063 10 mg + [^11C]T-773 | TAK-063 30 mg + [^11C]T-773 | TAK-063 100 mg + [^11C]T-773 | TAK-063 1000 mg + [^11C]T-773
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 2
liter/hour | 26.19 (1.099) | 18.31 (7.477) | 24.90 (2.209) | 88.86 (25.806) | 252.33 (21.971)

13. Secondary Outcome: Ratio of TAK-063 Metabolite Cmax to TAK-063 Cmax
Description: Cmax Ratio is the ratio of Cmax values of the metabolite compared to the parent calculated by dividing Cmax values of metabolite M-I with those of the parent drug TAK-063.
Time Frame: as for outcome 7
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | TAK-063 3 mg + [^11C]T-773 | TAK-063 10 mg + [^11C]T-773 | TAK-063 30 mg + [^11C]T-773 | TAK-063 100 mg + [^11C]T-773 | TAK-063 1000 mg + [^11C]T-773
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 2
ratio | 1.30 (0.271) | 0.83 (0.013) | 0.65 (0.361) | 0.99 (0.145) | 0.55 (0.001)

14. Secondary Outcome: Ratio of TAK-063 Metabolite M-I AUC( 0-24) to TAK-063 AUC (0-24)
Description: AUC Ratio is the ratio of AUC values of the metabolite compared to the parent calculated by dividing AUC values of metabolite M-I with those of the parent drug TAK-063.
Time Frame: as for outcome 7
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | TAK-063 3 mg + [^11C]T-773 | TAK-063 10 mg + [^11C]T-773 | TAK-063 30 mg + [^11C]T-773 | TAK-063 100 mg + [^11C]T-773 | TAK-063 1000 mg + [^11C]T-773
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 2
ratio | 0.93 (0.193) | 0.75 (0.064) | 0.66 (0.357) | 0.89 (0.199) | 0.54 (0.072)

15. Secondary Outcome: AUC During the Positron Emission Tomography (PET) Scan Period (AUC(Scan)) at 3 Hours Post-dose for TAK-063 and TAK-063 Metabolite M-I
Description: AUC values of TAK-063 and TAK-063 metabolite M-I during the PET scan at approximately 3 hours post TAK-063 administration.
Time Frame: 3 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | TAK-063 3 mg + [^11C]T-773 | TAK-063 10 mg + [^11C]T-773 | TAK-063 30 mg + [^11C]T-773 | TAK-063 100 mg + [^11C]T-773 | TAK-063 1000 mg + [^11C]T-773
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 2
ng*hr/mL
  TAK-063 | 9.51 (1.217) | 25.68 (0.970) | 63.18 (13.667) | 82.25 (16.404) | 269.32 (23.429)
  TAK-063 Metabolite M-I | 10.23 (3.850) | 22.56 (1.272) | 49.09 (21.273) | 85.13 (29.151) | 162.23 (6.527)

16. Secondary Outcome: Cavg During the Positron Emission Tomography (PET) Scan Period (AUC(Scan)) at 3 Hours Post-dose for TAK-063 and TAK-063 Metabolite M-I
Description: Cavg values of TAK-063 and TAK-063 metabolite M-I during the PET scan at approximately 3 hours post TAK-063 administration.
Time Frame: 3 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TAK-063 3 mg + [^11C]T-773 | TAK-063 10 mg + [^11C]T-773 | TAK-063 30 mg + [^11C]T-773 | TAK-063 100 mg + [^11C]T-773 | TAK-063 1000 mg + [^11C]T-773
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 2
ng/mL
  TAK-063 | 7.61 (0.974) | 20.54 (0.776) | 50.54 (10.934) | 65.80 (13.123) | 215.46 (18.743)
  TAK-063 Metabolite M-I | 8.18 (3.080) | 18.05 (1.018) | 39.27 (17.018) | 68.10 (23.321) | 129.78 (5.222)

17. Secondary Outcome: AUC During the Positron Emission Tomography (PET) Scan Period (AUC(Scan)) at 23 Hours Post-dose for TAK-063 and TAK-063 Metabolite M-I
Description: AUC values of TAK-063 and TAK-063 metabolite M-I during the PET scan at approximately 23 hours post TAK-063 administration. Data was not available for participants in the pilot cohort.
Time Frame: 23 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | TAK-063 3 mg + [^11C]T-773 | TAK-063 10 mg + [^11C]T-773 | TAK-063 30 mg + [^11C]T-773 | TAK-063 100 mg + [^11C]T-773
Number analyzed (Participants) | 2 | 2 | 1 | 3
ng*hr/mL
  TAK-063 | 1.75 (0.496) | 11.44 (4.243) | 21.22 (NA) — Standard deviation can not be calculated for 1 participant. | 21.15 (7.913)
  TAK-063 Metabolite M-I | 1.43 (0.071) | 8.20 (2.631) | 19.96 (NA) — Standard deviation can not be calculated for 1 participant. | 22.97 (15.919)

18. Secondary Outcome: Cavg During the Positron Emission Tomography (PET) Scan Period (AUC(Scan)) at 23 Hours Post-dose for TAK-063 and TAK-063 Metabolite M-I
Description: Cavg values of TAK-063 and TAK-063 metabolite M-I during the PET scan at approximately 23 hours post TAK-063 administration. Data is not available for the pilot cohort.
Time Frame: 23 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TAK-063 3 mg + [^11C]T-773 | TAK-063 10 mg + [^11C]T-773 | TAK-063 30 mg + [^11C]T-773 | TAK-063 100 mg + [^11C]T-773
Number analyzed (Participants) | 2 | 2 | 1 | 3
ng/mL
  TAK-063 | 1.40 (0.397) | 9.15 (3.394) | 16.97 (NA) — Standard deviation can not be calculated for 1 participant. | 16.92 (6.331)
  TAK-063 Metabolite M- | 1.15 (0.056) | 6.56 (2.105) | 15.97 (NA) — Standard deviation can not be calculated for 1 participant. | 18.37 (12.735)

ADVERSE EVENTS:
Time Frame: First dose of study drug to 30 days after last dose of study drug (up to 46 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | [^11C]T-773 | TAK-063
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 5/13 | 9/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | [^11C]T-773 (N=13) | TAK-063 (N=12)
Haematoma (Vascular disorders) | 0 | 4
Anxiety (Psychiatric disorders) | 1 | 2
Headache (Nervous system disorders) | 1 | 2
Infusion site pain (General disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
Tremor (Nervous system disorders) | 0 | 2
Catheter site pain (General disorders) | 1 | 1
Chest pain (General disorders) | 0 | 1
Claustrophobia (Psychiatric disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Infusion site erythema (General disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.